CLINICAL TRIAL: NCT00000738
Title: Randomized, Double-Blind, Placebo-Controlled Trial of Nimodipine for the Neurological Manifestations of HIV-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Miles (Industry); Glaxo Wellcome (Industry)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 162; 11137 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: AIDS Dementia Complex; HIV Infections
Keywords: Central Nervous System Diseases; Acquired Immunodeficiency Syndrome; AIDS Dementia Complex; AIDS-Related Complex; Zidovudine; Nimodipine
MeSH Terms: conditions — AIDS Dementia Complex; HIV Infections; Central Nervous System Diseases; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Nimodipine; Zidovudine

INTERVENTIONS:
Drug: Nimodipine
Drug: Zidovudine

SUMMARY:
PRIMARY: To assess the safety of nimodipine in the treatment of HIV-Associated Motor / Cognitive Complex (formerly AIDS dementia complex). To assess the systemic or central nervous system toxicities (e.g., rash, headache, gastrointestinal symptoms, nausea, dyspnea, muscle pain or cramp, acne) of nimodipine.

SECONDARY: To assess the efficacy of nimodipine in stabilizing the progression of HIV-Associated Motor / Cognitive Complex by improvement in neuropsychological test performance, peripheral neuropathy, or other neurologic manifestations.

HIV-infected patients may develop a condition known as HIV-Associated Motor / Cognitive Complex (also known as AIDS dementia complex) that causes damage to the nervous system, particularly the brain and spinal cord. Evidence exists that nimodipine protects nerve cells in culture from injury by HIV. Although nimodipine has been used in patients with other neurological problems, its safety and effectiveness in halting the progression of HIV-Associated Motor / Cognitive Complex is not yet known.

DETAILED DESCRIPTION:
HIV-infected patients may develop a condition known as HIV-Associated Motor / Cognitive Complex (also known as AIDS dementia complex) that causes damage to the nervous system, particularly the brain and spinal cord. Evidence exists that nimodipine protects nerve cells in culture from injury by HIV. Although nimodipine has been used in patients with other neurological problems, its safety and effectiveness in halting the progression of HIV-Associated Motor / Cognitive Complex is not yet known.

Forty patients currently taking zidovudine (AZT) or any other approved antiretroviral agent will be randomized to one of three treatment arms: high-dose nimodipine, low-dose nimodipine, or placebo. Additionally, six patients who are intolerant to standard antiretroviral therapy will be randomized to receive high- or low-dose nimodipine. Nimodipine is administered by mouth concurrently with patients' prestudy dose of antiretroviral agent. Treatment is given for 16 weeks, and patients are followed every 4 weeks. As an option, all patients may receive an additional 16 weeks of low-dose nimodipine.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Alternative or additional antiretroviral agents if on a stable dose for 8 weeks prior to study entry.
* Isoniazid.
* Anticonvulsants.
* Benzodiazepines and antidepressants (provided dose is stable prior to study entry).
* Symptomatic therapies (e.g., analgesics, antihistamines, antiemetics, and antidiarrheal agents).
* Maintenance therapy with clarithromycin, azithromycin, amikacin, ethambutol, clofazimine, ciprofloxacin, and rifampin for disseminated Mycobacterium avium infection.
* Maintenance therapy for opportunistic infections (e.g., PCP, MAI, CMV).

Patients must have:

* Documented HIV infection.
* HIV-Associated Motor / Cognitive Complex.
* Acceptable neurological and neuropsychological impairment scores.
* Estimated premorbid IQ of 70 or greater, consistent with completion of the sixth grade or ability to read at the sixth grade level. Current ability to read and comprehend a newspaper or history of such ability will satisfy this criterion for patients whose formal education stopped before the sixth grade. For patients who are illiterate, ability to make change from a dollar for a combined purchase of two items or the history of such ability will satisfy this criterion. In the absence of a functional definition, an age-correlated scaled score of > 5 on the Vocabulary Subtest of the WAIS-R or WISC-R may be used to establish IQ.
* Ability to provide written informed consent.

Prior Medication:

Required:

* AZT for at least 12 weeks prior to study entry or any other approved antiretroviral agent (i.e., ddI or ddC) for at least 8 weeks prior to study entry, except in antiretroviral-intolerant patients who must be off antiretrovirals for at least 4 weeks.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Active symptomatic AIDS-defining opportunistic infection (maintenance therapy for opportunistic infections, e.g., Pneumocystis carinii pneumonia, Mycobacterium avium infection, and cytomegalovirus, is permitted).
* Neoplasms other than basal cell carcinoma, in situ carcinoma of the cervix, or Kaposi's sarcoma without evidence of visceral involvement or that do not require systemic chemotherapy.
* Confounding neurological disorders, including the following:
* a) neurologic disease unrelated to HIV infection (such as multiple sclerosis, documented stroke, degenerative disease); b) chronic seizure disorders or head injuries if the condition results in functional impairment or is likely to interfere with evaluations; c) central nervous system (CNS) infections or neoplasms (such as toxoplasmosis, primary or metastatic CNS lymphoma, progressive multifocal leukoencephalopathy, cryptococcal or other fungal meningitis, tuberculous CNS infections, or untreated neurosyphilis).
* Severe premorbid psychiatric illness including bipolar illness, schizophrenia, and depression requiring electroconvulsive therapy.
* Major depression likely to interfere with evaluation or protocol compliance.

Concurrent Medication:

Excluded:

* Major psychotropic medication, including MAO inhibitors, phenothiazines, butyrophenones, barbiturates, or amphetamines (unless a stable dose is maintained for 30 days prior to study entry).
* Any ongoing maintenance therapy for confounding neurological disorders.

Patients with the following prior conditions are excluded:

Confounding neurological disorders defined in the "Exclusion Co-existing Conditions" field.

Prior Medication:

Excluded:

* Investigative drugs within 30 days prior to study entry.
* Confounding calcium channel antagonists (such as nifedipine, verapamil, diltiazem, and related drugs) within 4 weeks prior to study entry.

Active alcohol or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Study Completion 1994-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lipton S, Study Chair; Navia B, Study Chair; Simpson D, Study Chair; Tucker T, Study Chair
Locations (12):
- United States (12):
  - UCLA CARE Center CRS, Los Angeles, California
  - Northwestern University CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Bmc Actg Crs, Boston, Massachusetts
  - Beth Israel Deaconess - East Campus A0102 CRS, Boston, Massachusetts
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - Washington U CRS, St Louis, Missouri
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Case CRS, Cleveland, Ohio
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Background] Navia BA, Dafni U, Simpson D, Tucker T, Singer E, McArthur JC, Yiannoutsos C, Zaborski L, Lipton SA. A phase I/II trial of nimodipine for HIV-related neurologic complications. Neurology. 1998 Jul;51(1):221-8. doi: 10.1212/wnl.51.1.221. PMID 9674806
- [Background] Galgani S, Narciso P, Balestra P, Pigorini F, Pau F, Sette P, Tozzi V, Alba L, Grisetti S, Visco G. Nimodipine+ZDV vs ZDV in patients with ADC. Int Conf AIDS. 1994 Aug 7-12;10(1):205 (abstract no PB0248)